CLINICAL TRIAL: NCT06299540
Title: Benefits of an Individual Physical Activity Intervention on Health-related Quality of Life in Patients With Chronic Lymphocytic Leukemia Receiving Ibrutinib in Real-life Practice
Brief Title: Benefits of Individual Physical Activity Intervention on Health-related Quality of Life in Participants With Chronic Lymphocytic Leukemia
Acronym: QOLIBRI
Status: Recruiting | Type: Observational
Sponsor: Janssen Cilag S.A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: 54179060CLL4033; 54179060CLL4033 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Group 1: Individual Physical Activity Intervention: Participants with chronic lymphocytic leukemia (CLL) will be invited to perform physical activity according to a predefined intervention program. This program includes walking and weekly remote adapted physical activity sessions (2 sessions per week, the duration and difficulty of which will be adapted by the adapted physical activity [APA] trainer according to the Participant's abilities).
  Interventions: Behavioral: Individual Physical Activity Intervention (IPAI); Drug: Ibrutinib
- Group 2: Standard of Care: Participants with CLL will continue physical activity according to their lifestyle and the recommendations of the medical team.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Behavioral: Individual Physical Activity Intervention (IPAI) — No drug will be administered as a part of this study. The intervention will consist in an IPAI provided to participants for 6 months to practice physical activity in addition to their medical treatment in routine clinical practice settings. IPAI will be an adaptive program and will comprise two periods, the first period consisting in a supervised 4-month program and the second one in an unsupervised 2-month program to achieve greater autonomy.
  Groups: Group 1: Individual Physical Activity Intervention
Drug: Ibrutinib — No drug will be administered as a part of this study. Participants received ibrutinib as per their routine clinical practice settings.

SUMMARY:
The purpose of this study is to assess the impact of an individual physical activity intervention (IPAI) on health-related quality of life (HRQoL) in participants with first line or relapsed chronic lymphocytic leukemia (CLL) initiating ibrutinib in a routine clinical practice setting. HRQoL will be measured using functional assessment of cancer therapy - general scale (FACT-G).

ELIGIBILITY:
Inclusion Criteria:

* Participants newly treated with ibrutinib for first line or relapsed CLL (treatment is being initiated or has been initiated within the last 8 days as a maximum)
* Participants agreed to follow the individual physical activity intervention (IPAI)
* Participants using or having access to a compatible and appropriate electronic device such as smartphone, laptop or tablet
* Participants with Internet access at home and email address
* Participants agreed to wear a connected watch 24 hours a day for all the duration of the study

Exclusion Criteria:

* Pregnant participants or planning to become pregnant while enrolled in this study
* Participants with inability or deemed unsafe to practice physical activity
* Participants who have received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the inclusion visit
* Participants who are currently involved in an interventional study
* Participants with probable difficulties in using the digital tool autonomously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants aged at least 18 years of age with chronic lymphocytic leukemia (CLL).
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Health-related Quality of Life (HRQoL) by Using Functional Assessment of Cancer Therapy General (FACT-G) Total Score at Month 4.5 | Baseline and Month 4.5
  The FACT-G consists of 27 questions grouped in 4 dimensions: physical well-being (PWB; 7 items), social/family well-being (SWB; 7 items), emotional well-being (EWB; 6 items), and functional well-being (FWB; 7 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-G score is the summation of 4 subscale scores and ranges from 0-108. Higher scores for the scales and subscales indicate better HRQoL.

SECONDARY OUTCOMES:
Change from Baseline in HRQoL by Using Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) Total Score at Month 4.5, Month 6.5 and Month 12 | Baseline, Month 4.5, Month 6.5, and Month 12
  The FACT-Leu questionnaire consists of 44 questions grouped into 5 dimensions: PWB (7 items), SWB (7 items), EWB (6 items), FWB (7 items) and additional concerns (LEUS; 17 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-Leu score is the summation of 5 subscale scores and ranges from 0-176. Higher scores for the scales and subscales indicate better HRQoL.
Change from Month 4.5 in HRQoL by Using FACT-Leu Total Score at Month 6.5 | Month 4.5 and Month 6.5
  The FACT-Leu questionnaire consists of 44 questions grouped into 5 dimensions: PWB (7 items), SWB (7 items), EWB (6 items), FWB (7 items) and additional concerns (LEUS; 17 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-Leu score is the summation of 5 subscale scores and ranges from 0-176. Higher scores for the scales and subscales indicate better HRQoL.
Change from Month 6.5 in HRQoL by Using FACT-Leu Total Score at Month 12 | Month 6.5 and Month 12
  The FACT-Leu questionnaire consists of 44 questions grouped into 5 dimensions: PWB (7 items), SWB (7 items), EWB (6 items), FWB (7 items) and additional concerns (LEUS; 17 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-Leu score is the summation of 5 subscale scores and ranges from 0-176. Higher scores for the scales and subscales indicate better HRQoL.
Change from Baseline in HRQoL by Using Trial Outcome Index (TOI) Total Score at Month 4.5, Month 6.5, and Month 12 | Baseline, Month 4.5, Month 6.5, and Month 12
  The TOI questionnaire consists of 31 questions grouped into 5 dimensions: PWB (7 items), FWB (7 items) and additional concerns (LEUS; 17 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total TOI score is the summation of 5 subscale scores and ranges from 0-176. Higher scores for the scales and subscales indicate better HRQoL.
Change from Month 4.5 in HRQoL by Using Trial Outcome Index (TOI) Total Score at Month 6.5 | Month 4.5 and Month 6.5
  The TOI questionnaire consists of 31 questions grouped into 5 dimensions: PWB (7 items), FWB (7 items) and additional concerns (LEUS; 17 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total TOI score is the summation of 5 subscale scores and ranges from 0-176. Higher scores for the scales and subscales indicate better HRQoL.
Change from Month 6.5 in HRQoL by Using Trial Outcome Index (TOI) Total Score at Month 12 | Month 6.5 and Month 12
  The TOI questionnaire consists of 31 questions grouped into 5 dimensions: PWB (7 items), FWB (7 items) and additional concerns (LEUS; 17 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total TOI score is the summation of 5 subscale scores and ranges from 0-176. Higher scores for the scales and subscales indicate better HRQoL.
Change from Baseline in HRQoL by Using FACT-G Scale at Month 6.5 and Month 12 | Baseline, Month 6.5, and Month 12
  The FACT-G consists of 27 questions grouped in 4 dimensions: physical well-being (PWB; 7 items), social/family well-being (SWB; 7 items), emotional well-being (EWB; 6 items), and functional well-being (FWB; 7 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-G score is the summation of 4 subscale scores and ranges from 0-108. Higher scores for the scales and subscales indicate better HRQoL.
Change from Month 4.5 in HRQoL by Using FACT-G Scale at Month 6.5 | Month 4.5 and Month 6.5
  The FACT-G consists of 27 questions grouped in 4 dimensions: physical well-being (PWB; 7 items), social/family well-being (SWB; 7 items), emotional well-being (EWB; 6 items), and functional well-being (FWB; 7 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-G score is the summation of 4 subscale scores and ranges from 0-108. Higher scores for the scales and subscales indicate better HRQoL.
Change from Month 6.5 in HRQoL by Using FACT-G Scale at Month 12 | Month 6.5 and Month 12
  The FACT-G consists of 27 questions grouped in 4 dimensions: physical well-being (PWB; 7 items), social/family well-being (SWB; 7 items), emotional well-being (EWB; 6 items), and functional well-being (FWB; 7 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-G score is the summation of 4 subscale scores and ranges from 0-108. Higher scores for the scales and subscales indicate better HRQoL.
Percentage of Participants Achieving a Greater Than or Equal to (>=) 5-Point Improvement in the FACT-G Total Score at Months 4.5, 6.5, and 12 as Compared to Baseline | Baseline, Month 4.5, Month 6.5, and Month 12
  The FACT-G consists of 27 questions grouped in 4 dimensions: physical well-being (PWB; 7 items), social/family well-being (SWB; 7 items), emotional well-being (EWB; 6 items), and functional well-being (FWB; 7 items). Each item is given a weighted score of 0 to 4 and the score of each dimension are obtained by addition of the weighted scores of each item corresponding to the dimension. Total FACT-G score is the summation of 4 subscale scores and ranges from 0-108. Higher scores for the scales and subscales indicate better HRQoL.
Change from Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Total Score at Month 4.5, Month 6.5, and Month 12 | Baseline, Month 4.5, Month 6.5, and Month 12
  The FACIT-fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists of 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score is calculated as the sum of the 13 item scores (reserved scores [4 - score]) and ranges from 0 to 52, with a higher score indicating less fatigue. Positive changes from baseline indicate improvement of fatigue. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Change From Baseline in Total Sleep Time Using Connected Watch | Baseline, Month 4.5, Month 6.5, and Month 12
  Change from baseline in total sleep time (in hours) using connected watch will be assessed.
Change From Baseline in Total Sleep Score Using Connected Watch | Baseline, Month 4.5, Month 6.5, and Month 12
  Change from baseline in total sleep score (time asleep/time in bed) based on duration, regularity, depth and interruption using connected watch will be assessed.
Change From Baseline in Sleep Stages Using Connected Watch | Baseline, Month 4.5, Month 6.5, and Month 12
  Change from baseline in sleep stages (deep/light) using connected watch will be assessed.
Change From Baseline in Hospital Anxiety and Depression (HAD) Score at Month 4.5, Month 6.5, and Month 12 | Baseline, Month 4.5, Month 6.5, and Month 12
  The HAD scale is a 14-items measure that assesses anxiety and depressive disorders. The scale includes seven questions related to anxiety (total A) and seven others to the depressive dimension (total D). Each item is rated from 0 to 3. Two scores are derived from the scale, one related to anxiety and the other related to depression (maximum score for each score = 21). Higher scores indicate increased anxiety or depression.
Change From Baseline in Physical Fitness as Measured by Six-Minute Walk Test (6MWT) at Month 4.5, Month 6.5, and Month 12 | Baseline, Month 4.5, Month 6.5, and Month 12
  The 6MWT is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. It is easy to administer, better tolerated, and more reflective of activities of daily living than the other walk tests.
Change From Baseline in Physical Activity as Assessed by Number of Steps per Day Using Connected Watch | Baseline, Month 4.5, Month 6.5, and Month 12
  Change from baseline in physical activity as assessed by number of steps per day using connected watch will be reported.
Change From Baseline in Physical Activity as Assessed by the Number of Walking Sessions per Week using Connected Watch | Baseline, Month 4.5, Month 6.5, and Month 12
  Change from baseline in physical activity as assessed by the number of walking sessions per week using connected watch will be reported.
Change From Baseline in Physical Activity as Assessed by the Time of Walking Sessions per Week Using Connected Watch | Baseline, Month 4.5, Month 6.5, and Month 12
  Change from baseline in physical activity as assessed by the time of walking sessions per week using connected watch will be reported.
Change From Baseline in Physical Activity as Assessed by the Distance of Walking Sessions per Week Using Connected Watch | Baseline, Month 4.5, Month 6.5, and Month 12
  Change from baseline in physical activity as assessed by the distance of walking sessions per week using connected watch will be reported.
Percentage of Participants with Treatment-related Adverse Events | Up to 30 months
  Percentage of participants with treatment-related adverse events especially musculoskeletal and cardiovascular treatment-related adverse events will be reported.
Time to Treatment Discontinuation (TTD) | Months 6 and 12
  TTD is defined as the time between the first day of ibrutinib treatment and the day that ibrutinib is definitely stopped for whatever reason or death.
Reasons for Treatment Discontinuation | Up to Month 12
  Number of participants in each reason for treatment discontinuation will be reported. Reasons for treatment discontinuation are defined as: adverse events, lack of efficacy, patient's convenience, physician's decision, progression, death or other.
Percentage of Participants Who Still Wear the Connected Watch | Months 1, 3, 4.5, 6.5, and 12
  Percentage of participants who still wear the connected watch (adherence) will be assessed.
Percentage of Participants Retained by the Connected Watch (Start Wearing the Watch) | Months 1, 3, 4.5, 6.5, and 12
  Percentage of participants retained by the connected watch (start wearing the watch) will be assessed.
Percentage of Participants Agreed to Participate in the Study Among Eligible participants with Chronic Lymphocytic Leukemia (CLL) Initiation Ibrutinib Treatment | During the first 6 months (Feasibility period)
  Percentage of participants agreed to participate in the study among eligible participants with CLL initiation ibrutinib treatment will be reported.
For Group 1: Percentage of Participants Who Still Follow the Individual Physical Activity Intervention (IPAI) Among Those Who Have Started IPAI | Months 1, 3, 4.5, and 6.5
  Percentage of participants who still follow the IPAI among those who have started IPAI (Adherence) in group 1 will be assessed.
For Group 1: Percentage of Participants Who Follow the Adapted Physical Activity (APA) Sessions, the Walking Objectives and the APA Appointment as Scheduled With the APA Among Those Who Have Started IPAI | Months 1, 3, 4.5, and 4.6
  Percentage of participants who follow the adapted physical activity sessions, the walking objectives and the APA appointment as scheduled with the APA among those who have started IPAI (Compliance) in group 1 will be assessed.
For Group 1: Percentage of Participants Retained by the IPAI (First APA Videoconference Attended) Among Participants Enrolled in the Study | Months 1 and 3
  Percentage of participants retained by the IPAI (first APA videoconference attended) among participants enrolled in the study will be assessed.
For Group 1: Percentage of Participants who Completed the Supervised Period Among Participants Enrolled in the Study | Month 4.5
  Percentage of participants who completed the supervised period among participants enrolled in the study will be assessed.
For Group 1: Percentage of Participants who Completed the Unsupervised Period Among Participants Enrolled in the Study | Month 6.5
  Percentage of participants who completed the unsupervised period among participants enrolled in the study will be assessed.
For Group 1: Participant Satisfaction With the IPAI Measured With the Satisfaction Likert Scale | Months 4.5, 6.5, and 12
  Participant's' satisfaction will be assessed by Likert scales at Months 4.5 and 6.5 regarding coaching, proposed sessions, program content, program duration, impact on APA practice, overall satisfaction, willingness to continue and recommendation to others. Likert scales will assess participant's' satisfaction at Month 12 regarding impact on APA practice, overall satisfaction, willingness to continue and recommendation to others. Only one question is quantitative with score range from 0 (not at all satisfied) to 10 (totally satisfied) for global satisfaction. Participants are considered satisfied when score is greater than or equal to (>=) 6 and highly-satisfied when score is >=8. All other questions are qualitative and have 5-level Likert scales including: very satisfied, rather satisfied, neither satisfied nor dissatisfied, not really satisfied, not at all satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Cilag S.A.S., France Clinical Trial, Study Director — Janssen Cilag S.A.S.
Locations (1):
- Institut Universitaire du Cancer Toulouse Oncopole, Toulouse, France

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency